CLINICAL TRIAL: NCT00956800
Title: Remote Management of Diabetic Patients Via Data Transmission by Accu-Chek 360 Software
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbus Research Foundation (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Steven B. Leichter, M.D., Columbus Research Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Roche 360
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- telemedicine/study group (Experimental)
  Interventions: Other: Accu-Chek 360 software
- control group (Active Comparator)
  Interventions: Other: Normal care

INTERVENTIONS:
Other: Accu-Chek 360 software — Study group which will receive 3 routine office visits in the same time, and have two visits conducted by computer interaction, using the Accu-Chek 360 software.
  Arms: telemedicine/study group
Other: Normal care — Control group will receive 5 routine office visits in one year
  Arms: control group

SUMMARY:
The purpose of this study is to determine if providing some care to diabetic patients remotely, using Accuchek 360 yields at least the same clinical results for their diabetes care, according to existing guidelines, as providing all care to patients in person.

DETAILED DESCRIPTION:
This will be a non-inferiority study between two groups: a control group, which will receive 5 routine office visits in one year; and a study group which will receive 3 routine office visits in the same time, and have two visits conducted by computer interaction, using the Accuchek 360 software. All will be capable of independent care of their diabetes. All patients will be 19-65 years of age. The end-points will include similar changes in hemoglobin A1c, systolic and diastolic blood pressure, body mass index, lipid fractions, and similar levels of patient satisfaction with care.

There will be 50 patients in each group, matched for age and sex distribution, educational level, computer literacy, and type of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male and Female
* 19-65 years of age
* Type 1 and 2 diabetes
* Computer literate
* Independent care of diabetes
* Insulin pump allowed (Spirit pump only)
* Females on birth control
* Can demonstrate competency in the use of the Accuchek Aviva meter, reliability in doing regular home blood sugar determinations

Exclusion Criteria:

* Creatinine clearance < 30 cc/min
* Severe loss of vision (diabetic retinopathy)
* Severe diabetic neuropathy
* Known or suspected diabetic gastroparesis
* Patients with heart disease
* Patients with liver disease
* Drug or substantial alcohol use
* Use of pharmacological doses of glucocorticoids or other medications that affect blood sugar and blood pressure
* Females that are pregnant or are capable of becoming pregnant
* Insulin pump use other than Accucheck Spirit pump

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Columbus Research Foundation will take the objective data that constitutes the defined end-points of the study and enter it for each patient into an Access data base, using the established data base management system of Columbus Research Foundation. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven B Leichter, M.D., Principal Investigator — Endocrine Consultants
Locations (1):
- Columbus Research Foundation, Columbus, Georgia, United States